CLINICAL TRIAL: NCT00136383
Title: A Study of the Effects of Paroxetine vs. Duloxetine on Heart Rate Variability and Autonomic Cardiovascular Control
Brief Title: Comparing Paroxetine and Duloxetine on Cardiovascular Measures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00007207; 6956-05-3R0 (Other: DUMC)
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2007-09

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

INTERVENTIONS:
Drug: paroxetine versus duloxetine

SUMMARY:
This double-blind placebo-controlled trial is designed to test and to compare the cardiovascular profile of paroxetine controlled release (CR) with duloxetine in outpatients with depressive symptoms.

DETAILED DESCRIPTION:
This double-blind placebo-controlled study will test the hypothesis that greater reduction in heart rate variability will be associated with duloxetine than paroxetine in outpatients with major depressive disorder. We will also examine the relationship between changes in heart rate variability to the magnitude of serotonin and norepinephrine transporter occupancy produced by each drug.

ELIGIBILITY:
Inclusion Criteria:

* Depressive symptoms
* Ages 20-60
* In good medical health and not pregnant

Exclusion Criteria:

* Bipolar disorder
* Schizophrenia or other psychotic disorder
* Alcohol or other substance abuse within the last 3 months
* Cognitive impairment
* History of attempted suicide in the past 2 months and who score 4 or more on the suicide item of the MADRS

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
R-R interval change with deep breathing
Respiratory sinus arrhythmia

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS)
Hospital Anxiety and Depression Scale
Spielberger State-Trait Anxiety Inventory
Connor-Davidson Resilience Scale
Norepinephrine receptor occupancy
Serotonin receptor occupancy

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, M.D., Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States